CLINICAL TRIAL: NCT03960593
Title: Cohort of Patients> 70 Years Old With Cancer and / or Hematological Malignancy Treated With Chemotherapy and / or Immunotherapy and / or Targeted Therapy and / or New Generation Hormone Therapy After Oncogeriatric Evaluation and Therapeutic Revision on Public Assistance -Hospitals From Marseille
Brief Title: Cohort of Patients Over 70 Years of Age With Cancer and / or Hematological Malignancy
Acronym: ChimioAge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-56
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cancer and / or Hematological Malignancy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer and / or hematological: The population of the study will be all patients over 70 years of age with oncogeriatric HDJ cancer prior to initiation of oncologic therapy such as chemotherapy (oral or intravenous) and / or targeted therapy and / or immunotherapy and / or hormone therapy. new generation.
  Interventions: Other: Evaluation of the influence of geriatric factors

INTERVENTIONS:
Other: Evaluation of the influence of geriatric factors — Follow-up of patients> 70 years old with cancer pathologies to evaluate the influence of geriatric factors associated with a review of therapies on their care pathways and health conditions. We will be particularly interested in the main objective, the unplanned hospitalization rate at 3 months in patients> 70 years old with cancer treated in oncogeriatric HDJ before the initiation of oncological treatment such as chemotherapy (oral or intravenous) and / or targeted therapy and / or immunotherapy and / or new generation hormone therapy.

SUMMARY:
Follow-up of patients> 70 years old with cancer pathologies to evaluate the influence of geriatric factors associated with a review of therapies on their care pathways and health conditions. We will be particularly interested in the main objective, the unplanned hospitalization rate at 3 months in patients> 70 years old with cancer treated in oncogeriatric HDJ before the initiation of oncological treatment such as chemotherapy (oral or intravenous) and / or targeted therapy and / or immunotherapy and / or new generation hormone therapy.

DETAILED DESCRIPTION:
The aging of the French population is associated with a constant increase in the number of cancers in people over 75 years of age (1/3 of cancers diagnosed in patients ≥ 75 years).

Oncogeriatrics is a combination of two specialties, oncology and geriatrics. This practice aims to ensure that all elderly cancer patients are treated according to their condition through a multidisciplinary and multiprofessional approach. The improvement of the care of elderly people with cancer has been measured in Measure 23.4 of the 2009-2013 Cancer Plan. This objective is pursued through action 2.16 of the 2014-2019 Cancer Plan aimed at meeting the specific needs of elderly people with cancer, notably by relying on the organizational set-up of UCOGs (Coordination Units in Onco-Geriatrics). for an improvement of the management practices of this population and a structuring of clinical research in oncogeriatrics.

However, 85% of people over 75 have at least one pathology and more than 7 different molecules are delivered on average at least three times a year. Polypharmacy is a factor of frailty and the risk of functional decline is established from two prescribed drugs. Polypharmacy can be problematic in elderly patients with cancer who are treated with chemotherapy.

In our institution, we wanted to combine a review of therapies with this geriatric evaluation in elderly patients with cancer or haematological diseases managed by a systemic oncological treatment. In this context, during the evaluation sessions in day hospital (HDJ) of oncogeriatrics on the Assistance Publique-Hopitaux de Marseille (AP-HM), a medical assessment and a cross analysis between the usual treatments of patients (herbal medicine) and self-medication) and chemotherapy and / or immunotherapy and / or targeted therapy and / or new generation hormone therapy are routinely performed. The main objective of this work is to evaluate the influence of the therapeutic revisions associated with the EGS data on the unplanned hospitalization rate at 3 months and then the secondary objective of the impact on the course of treatment oncology, to become patients and their survival. For this purpose, we want to conduct a pilot observational cohort study, monocentric, prospective, descriptive for patients convened in oncogeriatric HDJ and each patient is followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 70 with an Oncoding score less than or equal to 14
* Patients receiving social security benefits
* suffering from cancerous pathology whatever the stage / grade and the associated comorbidities treated by chemotherapy and / or targeted therapy and / or immunotherapy and / or new generation hormone therapy
* Having read, understood and signed the non-opposition form

Exclusion Criteria:

* Patients refusing to participate in the research project
* Patients under guardianship or curatorship
* Patients who are not beneficiaries of a social security scheme

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population of the study will be all patients over 70 years of age with oncogeriatric HDJ cancer prior to initiation of oncologic therapy such as chemotherapy (oral or intravenous) and / or targeted therapy and / or immunotherapy and / or hormone therapy. new generation.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2024-05-06 (Estimated)

PRIMARY OUTCOMES:
Geriatric Assessment (EGS) on Geriatric HDJ | 3-6 moths
  Inclusion in HDJ and geriatric frailty collection (EGS) by the geriatrician in HDJ. Evaluation by pharmacist and collection in HDJ of the usual treatment, phytotherapy, future oncological treatment administered. Geriatric and pharmaceutical report in 24 hours sent to the treating physician and oncologist

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Couderc AL, Ninove L, Nouguerede E, Rey D, Rebroin M, Daumas A, Tomasini P, Greillier L, Salas S, Duffaud F, Dahan L, Duluc M, Garcia ME, Pluvy J, Chaleat S, Farnault L, Venton G, Fourie T, Nurtop E, de Lamballerie X, Villani P, Charrel R, Correard F. Acceptance, efficacy, and safety of COVID-19 vaccination in older patients with cancer. J Geriatr Oncol. 2022 Jul;13(6):850-855. doi: 10.1016/j.jgo.2022.05.002. Epub 2022 May 16. PMID 35589542